CLINICAL TRIAL: NCT00446368
Title: Phase II Study of RAD001 (Everolimus) in Patient's With Metastatic Renal Cell Cancer
Brief Title: Safety Study of RAD001 to Treat Patients With Metastatic Kidney Cancer
Acronym: RAD001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC IRB#03-0183-05; RCC-RAD-01 (Other: Novartis)
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: metastatic kidney cancer; metastatic renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): Subjects will take RAD001 (Everolimus) 10mg by mouth daily.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Participant will take RAD001 (Everolimus) 10mg by mouth once a day.
  Other Names: Everolimus

SUMMARY:
Patients with metastatic renal cell cancer will be enrolled to receive RAD001 to determine whether the use of RAD001 will result in an improvement in the time to tumor progression.

DETAILED DESCRIPTION:
Patients with metastatic renal cell cancer will be enrolled in the study if all eligibility criteria are met and they agree to participate. The participant will take RAD001 (Everolimus) 10mg by mouth once a day. During the first cycle, they will have blood work done once a week (4 weeks). On cycles thereafter they will have blood work on days 7 and 21. Once a month, the patient will have a chest x-ray. Every 8 weeks the patient will have a CT scan of the chest, abdomen and pelvis. If clinically indicated, additional tests will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have predominantly clear cell renal cancer (75%)
* Patients must have evidence of metastatic disease. Metastatic disease should not be progressing so as to require palliative treatment (e.g., radiation, surgery, etc), within 4 weeks of enrollment.
* Patients may have received no more than two prior regimens such as immunotherapy, chemotherapy or molecular targeted agents for renal cell carcinoma with at least 1 regimen consisting of a tyrosine kinase inhibitor (sorafenib or sunitinib). Four weeks must have elapsed from previous therapy.
* Patients must have adequate physiologic reserves as evidenced by lab values
* Effective birth control must be practiced by both male and female patients

Exclusion Criteria:

* Patients with central nervous system metastases are excluded, except those patients who have had complete excision or radiotherapy and remain asymptomatic, off steroids for 21 days, with no evidence of new disease as shown by MRI
* Patients known to be HIV positive are not eligible, although testing specifically for participation in this protocol is not required.
* Patients with a recent history of TIA (within 6 months), or are requiring regular antianginal therapy or are having claudication sufficient to limit activity are not eligible. Patients with a previous history of deep venous thrombosis or pulmonary embolism are not eligible.
* Patients with active autoimmune disease.
* Patients who have had steroid therapy within the past three weeks.
* Patients involving concurrent anticancer drug therapy. Any immunosuppressive drugs or any other experimental therapy.
* Female patients who are pregnant or lactating.
* The patient has an unstable medical condition, such as uncontrolled diabetes mellitus or hypertension; active infections requiring systemic antibiotics, antivirals, or antifungals; clinical evidence of cardiac or pulmonary dysfunction including, but not limited to: unstable CHF; uncontrolled arrhythmias; unstable coagulation disorders; or recent myocardial infarction (within 6 months).
* The patient has received any investigational agent(s) within 4 weeks of study entry.
* Patients with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count > 50,000 cells/mm3).
* Patients unable to maintain an absolute neutrophil count (ANC) of < 1,500 cells/mm3.
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the patient at unacceptable risk if he/she were to participate in the study.
* Prior malignancy (within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To collect data on time to tumor progression produced by the study treatment. | restaging every 8 weeks

SECONDARY OUTCOMES:
Response rate | restaging every 8 weeks
Duration of tumor response | restaging every 8 weeks
Safety and toxicity | AEs as occur
Six month and 12 month survival rate | at 6 months and at 12 months
Overall survival | restaging every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No